CLINICAL TRIAL: NCT05483166
Title: Engaging Parents in Neuropsychological Rehabilitation for Childhood Cancer Survivors: The "I'm Aware: Parents and Children Together" (ImPACT) Program - A Pilot Study
Brief Title: Engaging Parents in Neuropsychological Rehabilitation for Childhood Cancer Survivors: The ImPACT Program - A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Lisa Maria Wu, Associate Professor, University of Aarhus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ImPACT Child
Record Dates: First submitted 2022-07-19; First posted 2022-08-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Pediatric Cancer; Cognitive Dysfunction
Keywords: Pediatric Cancer; Cognitive Dysfunction; Neuropsychological Rehabilitation; Neurobehavioral Impairment
MeSH Terms: conditions — Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ImPACT program (Experimental): The ImPACT program consists of 8 weekly 1-hour sessions with homework between sessions.
  Interventions: Behavioral: ImPACT

INTERVENTIONS:
Behavioral: ImPACT — During the ImPACT program, the childhood cancer survivor and at least one parent collaborates on:
  1. Becoming aware of the child's core strengths and difficulties
  2. Helping the child to be optimally responsive to the guidance of the parent(s), and
  3. Creating compensatory strategies to respond to real-world manifestations of the child's difficulties and helping the child implement these strategies at home.

SUMMARY:
The aim of the present pilot study is to evaluate the feasibility, acceptability, and preliminary efficacy of a novel, context-sensitive neuropsychological rehabilitation intervention for childhood cancer survivors and their families.

DETAILED DESCRIPTION:
Cognitive impairment is the most common late effect in childhood cancer survivors, and despite the negative effects of these symptoms on quality of life, scholastic achievement and long-term socioeconomic outcomes, there continues to be no "gold standard" treatment for childhood cancer survivors with cognitive impairment.

Indeed, there is a dearth of research on interventions to treat cognitive impairment in childhood cancer survivors, and the relatively few studied interventions have proven limited effects. Arguably, four key elements are missing from a majority of studied interventions:1) transfer of learning to real-world functional outcomes, 2) awareness training to enhance compensatory strategy use, 3) inclusion of parents that could enhance transfer of learning to the home, and 4) recognition of the inter-related nature of cognitive, neurobehavioral, and psychological functions.

The "I'M aware: Parents and Children Together (ImPACT)" program is a novel, context-sensitive neuropsychological rehabilitation intervention that targets the above mentioned missing elements in previous rehabilitation efforts. The present pilot study aims to assess the feasibility, acceptability, and preliminary efficacy of this program in childhood cancer survivors with cognitive impairment in preparation for a large-scale randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Cancer diagnosis of a leukemia, lymphoma, or central nervous system tumor
* Completed primary treatment at least 6 months ago
* Not terminally ill
* Attend school
* Living with one or more parents who speak Danish and are willing to co-participate
* Screened as having parent-reported cognitive and/or neurobehavioral impairment

Exclusion Criteria:

• Confounding diagnosed or suspected psychiatric or medical condition unrelated to the cancer or its treatment that might contribute to cognitive or neurobehavioral impairment

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Parent-reported neurobehavioral functioning | Baseline (T1) to after last session (approximately 9 weeks later: Post-intervention, T3)
  The parent-report screening version of the Behavior Rating Inventory of Executive Function 2nd Edition (BRIEF-2). 12 items: answer format range: 1-3; total score range: 12-36. Higher score indicates more impairment.
Parent-reported cognitive functioning | Baseline (T1) to after last session (approximately 9 weeks later: Post-intervention, T3)
  The parent-report version of the Pediatric Perceived Cognitive Function (PedsPCF) Short Form. 7 items: answer format range 1-5; total score range: 7-35. Lower score indicates more impairment.

SECONDARY OUTCOMES:
Parent-reported neurobehavioral functioning | Baseline (T1) to 9 week after post-intervention (approximately 18 weeks later: Follow-up, T4)
  The parent-report version of the Behavior Rating Inventory of Executive Function 2nd Edition (BRIEF-2). 63 items: answer format range: 1-3; total score range: 63-189. Higher score indicates more impairment.
Parent-reported cognitive functioning | Baseline (T1) to 9 week after post-intervention (approximately 18 weeks later: Follow-up, T4)
  The parent-report version of the Pediatric Perceived Cognitive Function (PedsPCF) Short Form. 7 items: answer format range 1-5; total score range: 7-35. Lower score indicates more impairment.
Child-reported neurobehavioral functioning | Baseline (T1) to after last session (approximately 9 weeks later: Post-intervention, T3)
  The child-report version of the Behavior Rating Inventory of Executive Function 2nd Edition (BRIEF-2). 55 items: answer format range: 1-3; total score range: 55-165. Higher score indicates more impairment.
Child-reported neurobehavioral functioning | Baseline (T1) to 9 week after post-intervention (approximately 18 weeks later: Follow-up, T4)
  The child-report version of the Behavior Rating Inventory of Executive Function 2nd Edition (BRIEF-2). 55 items: answer format range: 1-3; total score range: 55-165. Higher score indicates more impairment.
Child-reported cognitive functioning | Baseline (T1) to after last session (approximately 9 weeks later: Post-intervention, T3)
  The child-report version of the Pediatric Perceived Cognitive Function (PedsPCF) Short Form. 7 items: answer format range 1-5; total score range: 7-35. Lower score indicates more impairment.
Child-reported cognitive functioning | Baseline (T1) to 9 week after post-intervention (approximately 18 weeks later: Follow-up, T4)
  The child-report version of the Pediatric Perceived Cognitive Function (PedsPCF) Short Form. 7 items: answer format range 1-5; total score range: 7-35. Lower score indicates more impairment.
Parent-reported pediatric quality of life | Baseline (T1) to after last session (approximately 9 weeks later: Post-intervention, T3)
  The parent-report version of the Pediatric Quality of Life (PedsQL) Core and Cancer scale. 23 items for the Core Scale, 25 items for the Cancer Scale: answer format range: 0-4; total score range: 0-100 (both scales). Lower scores indicate more impairment.
Parent-reported pediatric quality of life | Baseline (T1) to 9 week after post-intervention (approximately 18 weeks later: Follow-up, T4)
  The parent-report version of the Pediatric Quality of Life Inventory (PedsQL) Core and Cancer scale. 23 items for the Core Scale, 25 items for the Cancer Scale: answer format range: 0-4; total score range: 0-100 (both scales). Lower scores indicate lower quality of life.
Child-reported pediatric quality of life | Baseline (T1) to after last session (approximately 9 weeks later: Post-intervention, T3)
  The child-report version of the Pediatric Quality of Life (PedsQL) Core and Cancer scale. 23 items for the Core Scale, 25 items for the Cancer Scale: answer format range: 0-4; total score range: 0-100 (both scales). Lower scores indicate more impairment.
Child-reported pediatric quality of life | Baseline (T1) to 9 week after post-intervention (approximately 18 weeks later: Follow-up, T4)
  The child-report version of the Pediatric Quality of Life (PedsQL) Core and Cancer scale. 23 items for the Core Scale, 25 items for the Cancer Scale: answer format range: 0-4; total score range: 0-100 (both scales). Lower scores indicate more impairment.
Parent-reported pediatric anxiety and depression | Baseline (T1) to after last session (approximately 9 weeks later: Post-intervention, T3)
  The parent-report version of the Revised Children's Anxiety and Depression Scale (CADS) Short Form. 47 items: answer format range: 0-3; total score range: 0-27 (social phobia and panic disorder subscales), 0-30 (major depressive disorder subscale), 0-21 (social anxiety disorder subscale), 0-18 (generalized anxiety disorder and obsessive compulsive disorder subscales). Higher scores indicate more anxiety and depression.
Parent-reported pediatric anxiety and depression | Baseline (T1) to 9 week after post-intervention (approximately 18 weeks later: Follow-up, T4)
  The parent-report version of the Revised Children's Anxiety and Depression Scale (CADS) Short Form. 47 items: answer format range: 0-3; total score range: 0-27 (social phobia and panic disorder subscales), 0-30 (major depressive disorder subscale), 0-21 (social anxiety disorder subscale), 0-18 (generalized anxiety disorder and obsessive compulsive disorder subscales). Higher scores indicate more anxiety and depression.
Child-reported pediatric anxiety and depression | Baseline (T1) to after last session (approximately 9 weeks later: Post-intervention, T3)
  The child-report version of the Revised Children's Anxiety and Depression Scale (CADS) Short Form. 47 items: answer format range: 0-3; total score range: 0-27 (social phobia and panic disorder subscales), 0-30 (major depressive disorder subscale), 0-21 (social anxiety disorder subscale), 0-18 (generalized anxiety disorder and obsessive compulsive disorder subscales). Higher scores indicate more anxiety and depression.
Child-reported pediatric anxiety and depression | Baseline (T1) to 9 week after post-intervention (approximately 18 weeks later: Follow-up, T4)
  The child-report version of the Revised Children's Anxiety and Depression Scale (CADS) Short Form. 47 items: answer format range: 0-3; total score range: 0-27 (social phobia and panic disorder subscales), 0-30 (major depressive disorder subscale), 0-21 (social anxiety disorder subscale), 0-18 (generalized anxiety disorder and obsessive compulsive disorder subscales). Higher scores indicate more anxiety and depression.
Parent-reported pediatric fatigue | Baseline (T1) to after last session (approximately 9 weeks later: Post-intervention, T3)
  The parent-report version of the Pediatric Quality of Life - Multidimensional Fatigue Scale (PedsQL-MFS). 18 items: answer format range 0-4; total score range: 0-100. Lower score indicates more fatigue.
Parent-reported pediatric fatigue | Baseline (T1) to 9 week after post-intervention (approximately 18 weeks later: Follow-up, T4)
  The parent-report version of the Pediatric Quality of Life - Multidimensional Fatigue Scale (PedsQL-MFS). 18 items: answer format range 0-4; total score range: 0-100. Lower score indicates more fatigue.
Child-reported pediatric fatigue | Baseline (T1) to after last session (approximately 9 weeks later: Post-intervention, T3)
  The child-report version of the Pediatric Quality of Life - Multidimensional Fatigue Scale (PedsQL-MFS). 18 items: answer format range 0-4; total score range: 0-100. Lower score indicates more fatigue.
Child-reported pediatric fatigue | Baseline (T1) to 9 week after post-intervention (approximately 18 weeks later: Follow-up, T4)
  The child-report version of the Pediatric Quality of Life - Multidimensional Fatigue Scale (PedsQL-MFS). 18 items: answer format range 0-4; total score range: 0-100. Lower score indicates more fatigue.
Parent sense of competence | Baseline (T1) to after last session (approximately 9 weeks later: Post-intervention, T3)
  The Parenting Sense of Competence Scale (PSC scale).17 items: answer format range 1-6; total score range: 16-102. Higher score indicates more competence.
Parent sense of competence | Baseline (T1) to 9 week after post-intervention (approximately 18 weeks later: Follow-up, T4)
  The Parenting Sense of Competence Scale (PSC scale). 17 items: answer format range 1-6; total score range: 16-102. Higher score indicates more competence.
Parent-reported participant motivation | After last session (approximately 9 weeks after Baseline assessment (T1): Post-intervention, T3)
  The 7-item interest/enjoyment subscale of the Intrinsic Motivation Inventory (IMI). 7 items: answer format range 1-7; total score range: 1-7. Higher score indicates more motivation.
Child-reported participant motivation | After last session (approximately 9 weeks after Baseline assessment (T1): Post-intervention, T3))
  The 7-item interest/enjoyment subscale of the Intrinsic Motivation Inventory (IMI). 7 items: answer format range 1-7; total score range: 1-7. Higher score indicates more motivation.
Parent-reported participant satisfaction | After last session (approximately 9 weeks after Baseline assessment (T1): Post-intervention, T3)
  The Client Satisfaction Questionnaire (CSQ-8). 8 items: answer format range 1-4; total score range: 8-32. Higher score indicates better satisfaction.
Child-reported participant satisfaction | After last session (approximately 9 weeks after Baseline assessment (T1): Post-intervention, T3)
  The Client Satisfaction Questionnaire (CSQ-8). 8 items: answer format range 1-4; total score range: 8-32. Higher score indicates better satisfaction.
Objective cognitive functioning (Child only) | Baseline (T1) to after last session (approximately 9 weeks later: Post-intervention, T3)
  Standard neuropsychological test battery. Different scoring formats.
Objective cognitive functioning (Child only) | Baseline (T1) to 9 week after post-intervention (approximately 18 weeks later: Follow-up, T4)
  Standard neuropsychological test battery. Different scoring formats.

OTHER OUTCOMES:
Qualitative Interviews | 9 week after post-intervention (approximately 18 weeks after Baseline assessment (T1): Follow-up, T4)
  Following the T4 assessment, the child and parent(s) will be invited to participate in a 30-minutes semi-structured, audio recorded interview.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Wu, PhD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No